CLINICAL TRIAL: NCT03169348
Title: The Effect of Direct Antiviral Therapy on Hepatitis c Virus-related Thrombocytopenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCV
Record Dates: First submitted 2017-05-25; First posted 2017-05-30 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Experimental): Hepatitis- C virus with thrombocytopenia
  Interventions: Drug: sofosbuvir daclatasvir; Drug: Ledipasvir/sofosbuvir

INTERVENTIONS:
Drug: sofosbuvir daclatasvir — oral tablets
Drug: Ledipasvir/sofosbuvir — oral tablets

SUMMARY:
Autoimmune thrombocytopenic purpura is an immunological disorder characterized by increased platelet destruction due to presence of anti-platelet antibodies. Hepatitis C virus infection, which is one of the most common chronic viral infections worldwide, may cause secondary chronic immune thrombocytopenic purpura. It seemed to play a pathogenic role in autoimmune thrombocytopenic purpura. Moreover, the successful response (negative hepatitis C virus - ribonucleic acid) to tapered steroids and antiviral therapy was useful to revert thrombocytopenia

ELIGIBILITY:
Inclusion Criteria:

* Hepatitis C virus infection and thrombocytopenia before treatment

Exclusion Criteria:

* Infection Hepatitis B virus
* Hypersplenism
* Diseases affecting Bone marrow
* Major clotting factors abnormalities eg. Disseminated intravascular coagulopathy, severe Prothrombin deficiency

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
the mean difference on the platelet count | 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No